CLINICAL TRIAL: NCT03309280
Title: Influence of Different Parameters on Extubation Time After Cardiac Surgery.
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, FAHA, Head of Department, Astes
Other Study IDs: VACC Study
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient at risk for OSA scheduled for Cardiac surgery: Patients with a positive STOP-Bang and DES-OSA score (that means patients at risk for OSA)
  Interventions: Other: Duration of intubation; Diagnostic Test: Evolution of the renal function
- Patient not at risk for OSA scheduled for Cardiac surgery: Patients with a negative STOP-Bang and DES-OSA score (that means patients not at risk for OSA)
  Interventions: Other: Duration of intubation; Diagnostic Test: Evolution of the renal function

INTERVENTIONS:
Other: Duration of intubation — Time between intubation in the operating room and exhumation in the Intensive Care Unit.
Diagnostic Test: Evolution of the renal function — Evolution of the renal function in the next two days

SUMMARY:
The aim of this study is to determine which factors could be at risk of delayed extubation after cardiac surgery.

DETAILED DESCRIPTION:
The aim of this study is to determine which factors could be at risk of delayed extubation after cardiac surgery. Several parameters of ventilation and infusion were recorded during surgery. A statistical analysis will be performed to determine if one of many of these are significant. The investigator does not assign specific interventions to the study participants, so the present study is observational and not interventional.

ELIGIBILITY:
Inclusion Criteria:

* All patients for elective cardiac surgery

Exclusion Criteria:

* Emergency procedures

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for cardiac surgery in the Saint-Luc Bouge hospital.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Time of extubation | 2 Days
  Time when extubation is performed

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deflandre, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc de Bouge, Bouge, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No